CLINICAL TRIAL: NCT02421627
Title: Study on the Mechanism of Moxibustion Effect on Treating Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: Moxibustion for Diarrhea-predominant Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYS2015-01
Record Dates: First submitted 2015-04-08; First posted 2015-04-20 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2019-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: moxibustion; irritable bowel syndrome; Magnetic Resonance Imaging
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxibustion group (Experimental): Receiving moxibustion treatment
  Interventions: Device: moxibustion
- Sham moxibustion group (Sham Comparator): Receiving sham moxibustion.
  Interventions: Device: Sham moxibustion

INTERVENTIONS:
Device: moxibustion — Acupoints: Tianshu (ST25，bilateral), Zusanli (ST36，bilateral). using mild-warm moxibustion，the surface temperature of acupoints were maintained at 43 ℃ ± 1 ℃, 30min for each acupoint, once every other day, three times a week, a total of six weeks treatment. After the treatment, subjects were followed up at weeks 12, 18 and 24.
  Arms: Moxibustion group
Device: Sham moxibustion — Acupoints: Tianshu (ST25，bilateral), Zusanli (ST36，bilateral); using sham mild-warm moxibustion，the surface temperature of acupoints were maintained at 37 ℃ ± 1 ℃, 30min for each acupoint, once every other day, three times a week, a total of six weeks treatment. After the treatment, subjects were followed up at weeks 12, 18 and 24.
  Arms: Sham moxibustion group

SUMMARY:
To observe the safety and efficacy of moxibustion on diarrhea-predominant irritable bowel syndrome and evaluation by Magnetic Resonance Imaging (MRI), Event related potential (ERP).

DETAILED DESCRIPTION:
1. A randomized controlled trial
2. Moxibustion treatment, sham control
3. To observe the safety and efficacy of moxibustion treatment versus placebo control
4. Evaluation by intestinal microbial structural and diversity changes using 16S rDNA sequencing
5. Evaluation by structural MRI and resting state-functional MRI
6. Evaluation by ERP

ELIGIBILITY:
Inclusion Criteria:

1. Diarrhea-predominant IBS patients who met the Rome III diagnostic criteria;
2. Age 18-65 years old, male or female;
3. Volunteered for the trial, signed the informed consent

Exclusion Criteria:

1. Intestinal organic disease;
2. Constipation-predominant IBS;
3. Alternating diarrhea and constipation IBS;
4. Unstructured IBS;
5. At the same time, application of smecta, dicetel, cisapride or traditional Chinese medicine;
6. Combined liver, kidney, heart or mental disease patients;
7. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Total efficacy (Adequate relief responder) | Week 6
  The ratio of the number of responders and the total number of participants in each group. Adequate relief responder is the participant who considered effective treatment in the self-assessment.

SECONDARY OUTCOMES:
Total efficacy (Adequate relief responder) | Week 12, 18 and 24
  Differences in Adequate relief responder between groups
Symptom severity score (SSS) | Week 6, 12, 18 and 24
  Differences in the mean changes of SSS score from baseline between groups
The proportion of responder to SSS | Week 6, 12, 18 and 24
  The differences of the proportion of responders between groups. Defined the SSS score decreased more than 50 points from baseline as responder.
Bristol stool form scale (BSS) | Week 6, 12, 18 and 24
  Differences in the mean changes of BSS score from baseline between groups
Quality of life questionnaire (IBS-QOL) | Week 6
  Differences in the mean changes of IBS-QOL score from baseline between groups
hospital anxiety and depression score (HADS) | Week 6
  Differences in the mean changes of HADS score from baseline between groups
Self-rating anxiety scale (SAS) | Week 6
  Differences in the mean changes of SAS score from baseline between groups
Self-rating Depression Scale (SDS) | Week 6
  Differences in the mean changes of SDS score from baseline between groups
Diarrhea frequency per day | Week 6, 12, 18 and 24
  Differences in the mean changes of Diarrhea frequency per day from baseline between groups
Urgency of defecation | Week 6, 12, 18 and 24
  Differences in the mean changes of Urgency of defecation from baseline
Safety evaluation (Number of participants with treatment-related adverse events as assessed by CTCAE v4.0) | Week 6, 12, 18 and 24
  Eg.moxibustion related burns, blistering, etc

OTHER OUTCOMES:
Brain structures （gray matter, white matter）MRI | Week 6
resting-state functional MRI | Week 6
  Analysis with methods of regional homogeneity，ALFF/fALFF，functional connectivity.
Magnetic Resonance Spectroscopy (MRS) | Week 6
  The ratio of glutamate complex (Glx) peak area and creatine ratio (Cr) of the cingulate cortex and insula.
Event-related potentials (ERP) | Week 6
  Measurement of brain resting state energy atlas and the amplitude changes of each major components during the task and latency.
Intestinal microbiota changes | Week 6
  Fecal microbial structural and diversity changes
Brain-gut microbiota interaction | Week 6
  Multiple regression analysis to establish the association between intestinal microbiota and brain

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, MD,PhD, Study Chair — Shanghai University of TCM
Locations (3):
- China (3):
  - Shanghai Institute of Acupuncture, Moxibustion and Meridian, Shanghai, Shanghai Municipality
  - Shanghai Traditional Chinese Medicine-Integrated Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Yueyang Integrated Chinese and Western Medicine Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Bao C, Wu L, Shi Y, Shi Z, Jin X, Shen J, Li J, Hu Z, Chen J, Zeng X, Zhang W, Ma Z, Weng Z, Li J, Liu H, Wu H. Long-term effect of moxibustion on irritable bowel syndrome with diarrhea: a randomized clinical trial. Therap Adv Gastroenterol. 2022 Feb 23;15:17562848221075131. doi: 10.1177/17562848221075131. eCollection 2022. PMID 35222693
- [Derived] Bao C, Zhang J, Liu J, Liu H, Wu L, Shi Y, Li J, Hu Z, Dong Y, Wang S, Zeng X, Wu H. Moxibustion treatment for diarrhea-predominant irritable bowel syndrome: study protocol for a randomized controlled trial. BMC Complement Altern Med. 2016 Oct 24;16(1):408. doi: 10.1186/s12906-016-1386-4. PMID 27776494